CLINICAL TRIAL: NCT04536311
Title: Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Brief Title: Surgical Stabilization of Rib Fractures While Awake or Under Appropriate Sedation by Paravertebral Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Weigang Zhao, Clinical Professor, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-036-(1)
Record Dates: First submitted 2020-08-07; First posted 2020-09-02 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Rib Fracture Multiple; Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paravertebral block in surgical stabilization of rib fractures under awake or appropriate sedation (Experimental): patients receive internal fixation for multiple rib fractures using paravertebral nerve block anesthesia in awareness status and keep spontaneous breath
  Interventions: Procedure: internal fixation of mulitiple rib fracture

INTERVENTIONS:
Procedure: internal fixation of mulitiple rib fracture — The dislocated rib fracture was anatomically reduced, and then fixed with appropriate equipment to prevent the fracture from being displaced again

SUMMARY:
Tracheal intubation and general anesthesia has been considered a safe and conventional routine methodology for thoracic surgery, include multiple rib fratcure. However,adverse effects such as sore throat, pain, hoarseness, and respiratory complications are common after that. In this study, we decide to perform surgical stabiliazation of rib fractures by paravertebral block surgical stabiliazation of rib fractures under awake or appropriate sedation without endotracheal intubation keeping spontaneous respiration to investigate its safety and feasibility.

DETAILED DESCRIPTION:
Rib fracture is common in the world,especially in chest trauma. Conservative treatment is used to it for many years but the effect is not well because of continuous pain caused by the dislocation of broken rib. Surgical stabiliazation of rib fractures can relieve the pain rapidly and help patient recover to work early. This kind of surgery is constantly conducted with tracheal intubation and general anesthesia. However,adverse effects such as sore throat, pain, hoarseness, and respiratory complications are common after that. So we think perform surgical stabiliazation of rib fractures under awake or appropriate sedation without endotracheal intubation keeping spontaneous respiration to investigate its safety and feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Simple rib fracutures patients
* No other truama
* Unilatieral rib fractures
* Total number of rib fractures is less than 5
* At least one rib dislocation
* 18-80 years old
* ASA grade I-II
* BMI<30
* Preoperative arterial partial pressure of oxygen > 60mmhg
* Partial pressure of carbon dioxide < 50mmhg

Exclusion Criteria:

* Difficult airway
* History of esophageal reflux
* Myasthenia gravis
* Coagulation disorders
* Gastrointestinal ulcer
* Gastrointestinal bleeding
* Anesthetic drugs allergy history
* Asthma
* Chronic obstructive pulmonary disease
* Pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
conversion to tracheal intubation | during surgery
  index of consciousness(IOC): If the scale low zhan 40 or high than 60, it need intubation
pain score | 6 hours after operation
  Numerical Rating Scale(NRS): 0-10 is used to represent different degrees of pain, 0 is painless and 10 is severe pain. The grading criteria of pain were: 0: no pain; 1-3: mild pain; 4-6: moderate pain; 7-10: severe pain
pain score | 12 hours after operation
  Numerical Rating Scale(NRS): 0-10 is used to represent different degrees of pain, 0 is painless and 10 is severe pain. The grading criteria of pain were: 0: no pain; 1-3: mild pain; 4-6: moderate pain; 7-10: severe pain
pain score | 24 hours after operation
  Numerical Rating Scale(NRS): 0-10 is used to represent different degrees of pain, 0 is painless and 10 is severe pain. The grading criteria of pain were: 0: no pain; 1-3: mild pain; 4-6: moderate pain; 7-10: severe pain

SECONDARY OUTCOMES:
operation time | during surgery
  operation time
blood loss | during surgery
  blood loss
days of stay hospital | from the date of hospitalization to the date of leave hospital,assessed up to 100 months
  days of stay hospital
costs of stay hospital | from the date of hospitalization to the date of leave hospital,assessed up to 100 months
  costs of stay hospital
PONV score | 6 hours after operation
  Visual analogue scale (VAS). 1-10 is used to represent different degrees of nausea and vomiting. 1 ~ 4 was mild, 5 ~ 6 was moderate, 7 ~ 10 was severe
PONV score | 12 hours after operation
  Visual analogue scale (VAS). 1-10 is used to represent different degrees of nausea and vomiting. 1 ~ 4 was mild, 5 ~ 6 was moderate, 7 ~ 10 was severe
PONV score | 24 hours after operation
  Visual analogue scale (VAS). 1-10 is used to represent different degrees of nausea and vomiting. 1 ~ 4 was mild, 5 ~ 6 was moderate, 7 ~ 10 was severe

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yang, Study Chair — Shanghai Jiao Tong University affiliated 6th people's hospital
Locations (1):
- Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wu W, Gao X, Liu P, Zhao W, Yang Y. Paravertebral block analgesia during surgical stabilization for rib fractures patients under conscious state: a single-arm, pilot study and post-hoc analysis. J Cardiothorac Surg. 2025 Mar 21;20(1):161. doi: 10.1186/s13019-025-03397-8. PMID 40119455